CLINICAL TRIAL: NCT01026909
Title: Intraarticular Corticosteroid Therapy in Legg-Calve Perthes Disease: a Randomized Controlled Clinical Trial.
Brief Title: Intraarticular Corticosteroid Therapy in Perthes Disease.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Klane White, Assitant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEF-24812
Record Dates: First submitted 2009-10-06; First posted 2009-12-07 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Legg-Calve Perthes Disease
MeSH Terms: conditions — Legg-Calve-Perthes Disease | interventions — triamcinolone hexacetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Injection (Experimental): Patients in this arm receive one single dose of Triamcinolone hexacetonide injectable suspension (Aristopan), USP, 20mg/mL Parenteral. They will aso be enrolled in physical therapy.
  Interventions: Drug: Aristospan 20mg
- Control (No Intervention): Patients will be enrolled in physical therapy

INTERVENTIONS:
Drug: Aristospan 20mg — Triamcinolone hexacetonide injectable suspension, USP, 20mg/mL Parenteral. One single dose.
  Arms: Injection

SUMMARY:
Legg-Calve-Perthes disease (LCP) represents the loss of blood flow to the head of the femur, resulting in significant hip pain and potential long term disability. This study represents a single center, randomized, prospective, controlled study comparing the treatment of LCP with an intraarticular corticosteroid (triamcinolone hexacetonide) injection with traditional nonoperative treatment.

DETAILED DESCRIPTION:
Legg-Calve-Perthes disease (LCP) represents the loss of blood flow to the head of the femur, resulting in significant hip pain and potential long term disability. The cause of LCP is still unknown, but tends to occur predominantly in boys from ages 4-12. For the majority of those affected, observation and symptomatic treatment with oral antiinflammatories, such as ibuprofen, is indicated. This study represents a single center, randomized, prospective, controlled study comparing the treatment of LCP with an intraarticular corticosteroid (triamcinolone hexacetonide) injection with traditional nonoperative treatment. The investigators will test for improved outcomes by measuring functional outcomes (PODCI and ASKp questionnaires, StepWatch activity monitor), hip range of motion and visual-analog pain scales. The investigators hypothesize that injections of corticosteroids (potent, injectable antiinflammatories) will result in improved overall function through decreased pain and increased hip range of motion in this patient population.Additional biological research will be performed. There is no human information on the inflammatory response that occurs in the hip joint of children with Perthes disease, and there are no true animal models of Perthes disease. To better understand the pathobiology of Perthes disease, the collection of joint fluid from both hips may provide insight into the treatment of a disease for which we currently have no explanation of cause, and consequently no therapies

ELIGIBILITY:
Inclusion Criteria:

* age of 4 to 12 years
* diagnosed with Idiopathic osteonecrosis of the femoral head
* symptoms less than 12 months old.

Exclusion Criteria:

* Symptoms for more than 12 months
* Previous treatment other than anti-inflammatories, crutches or bed rest
* Subjects more than 8 years old or have a hand bone age greater than 6 years old and lateral pillar B or B/C disease.
* Bilateral hip disease
* Personal or family history of problems with general anesthesia
* Prior steroid treatment
* Previous diagnosis of:

  * Asthma
  * Identifiable rheumatologic condition
  * Metabolic Diseases (including but not limited to Gaucher's disease or congenital hypothyroidism)
  * Sickle cell disease
  * Known pain syndrome
  * Hip sepsis
  * Prior malignancy (solid organ or bone marrow transplant)
  * Blood Clotting disorder

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2009-03; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klane K White, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Observation
Period: Overall Study
Arm/Group | Injection | Control
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Injection | Control | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (0) | 7.33 (2.08) | 7.33 (2.08)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Variable: Function. The Pediatric Outcomes Data Collection Instrument (PODCI) Will be the Primary Endpoint as a Measure of Function and Health Related Quality of Life at 12 Months Post Injection.
Description: The Pediatric Outcomes Data Collection Instrument (PODCI) is designed to be completed by the parent/guardian of a child ten years of age or younger who has knowledge of the child's conditions. The eight scales generated from these instruments are:
  Upper Extremity and Physical Function Scale; Transfer and Basic Mobility Scale; Sports/Physical Functioning Scale; Pain/Comfort; Treatment Expectations Scale; Happiness Scale; Satisfaction with Symptoms Scale and Global Functioning Scale. The results of each scale are standardized into a scale of 0-100 where 0 indicates the worst outcome and 100 the best.
  We decided to report Global Functioning only due to space limitations. Also the Global Functioning scale encompasses items from other scales.
Time Frame: This exam is to be administered at time of enrollment and at 4 and 12 months follow up visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injection | Control
Number analyzed (Participants) | 1 | 2
units on a scale
  After Treatment (12 months) Global Functioning Sca | 97 | 97.5 (3.53)
  Before treatment - Global Functioning Scale | 64 | 79 (2.83)

2. Secondary Outcome: Second Outcome Variable: Ambulatory Activity. It Will be Defined as Average Steps/Day as Measured by the StepWatch Activity Monitor for a 7 Day Sample.
Time Frame: StepWatch monitor will be used 7 days prior to treatment and 4 weeks, 4 months and 12 months follow up visits
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Injection | Control
Number analyzed (Participants) | 1 | 2
steps/day
  Baseline- Average Number of steps per day | 6287 | 1448.04 (1873.78)
  4 weeks Follow Up- Average Number of steps per d | 1782.19 | 2521.91 (1046.12)
  4 months follow up- average # of steps per day | 6985.89 | 2687.57 (1999.4)
  12 months follow up- average # of steps per day | 6990 | 2158.7 (865.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Injection | Control
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes